CLINICAL TRIAL: NCT03147716
Title: Effectiveness Trial of Methods for Engaging Parents Into Parenting Interventions
Brief Title: Parent Engagement Package: Comparing Strategies for Engaging Parents Into Parenting Programs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Mesa Public Schools (Unknown)
Responsible Party: Principal Investigator, Emily Winslow PhD, Assistant Research Professor, Arizona State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY00001365; R01DA033352 (NIH)
Record Dates: First submitted 2017-04-17; First posted 2017-05-10 (Actual); Last update posted 2019-08-09 (Actual); Status verified 2019-08

CONDITIONS: Patient Compliance
MeSH Terms: conditions — Patient Compliance

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to one of five conditions: 1) enrollment flyer only; 2) enrollment flyer + testimonial booklet; 3) enrollment flyer + teacher endorsement; 4) enrollment flyer + provider engagement call; or 5) all four engagement strategies.
Who Masked: Participant
Masking Description: single-blind masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Enrollment Flyer (Active Comparator): Participants in this condition received one of the strategies in the Parent Engagement Package: an enrollment flyer that provided information about the Triple P Positive Parenting Program being offered at their child's school, including the location of meetings, free childcare, topics covered, choice of days/times and English or Spanish groups, and an enrollment form. Parents who returned the enrollment form received automated text, email and/or phone reminders and a confirmation letter prior to each parenting program session.
  Interventions: Other: Enrollment Flyer
- Enrollment Flyer & Testimonial Booklet (Experimental): Participants in this condition received two of the strategies in the Parent Engagement Package: the enrollment flyer plus a two-page, testimonial booklet that included photos and quotes from parents and children describing benefits other parents reported after participating in the Triple P Positive Parenting Program and fun activities children reported about the childcare. The booklet also contained the location of meetings, free childcare, choice of days/times and English or Spanish groups, and an enrollment form.
  Interventions: Other: Enrollment Flyer; Other: Testimonial Booklet
- Enrollment Flyer & Teacher Endorsement (Experimental): Participants in this condition received two of the strategies in the Parent Engagement Package: the enrollment flyer plus a teacher endorsement of the Triple P Positive Parenting Program. The teacher also gave the participant a colorful brochure that included information about the location of meetings, free childcare, topics covered, choice of days/times and English or Spanish groups, and an enrollment form.
  Interventions: Other: Enrollment Flyer; Other: Teacher Endorsement
- Enrollment Flyer & Engagement Call (Experimental): Participants in this condition received two of the strategies in the Parent Engagement Package: the enrollment flyer plus an engagement call from a Triple P provider. Providers followed a manualized protocol for implementing the engagement call, which included strategies to increase parental motivation to participate in Triple P and reduce barriers to participation.
  Interventions: Other: Enrollment Flyer; Other: Provider Engagement Call
- All Engagement Strategies (Experimental): Participants in this condition received all engagement strategies in the Parent Engagement Package: enrollment flyer, testimonial booklet, teacher endorsement, and provider engagement call.
  Interventions: Other: Enrollment Flyer; Other: Testimonial Booklet; Other: Teacher Endorsement; Other: Provider Engagement Call

INTERVENTIONS:
Other: Enrollment Flyer — Enrollment flyer that provided information about the Triple P Positive Parenting Program and an enrollment form.
Other: Testimonial Booklet — Booklet that included quotes and photos from parents who had previously participated in the Triple P Positive Parenting Program and/or their children who participated in the free childcare, as well as an enrollment form.
  Arms: All Engagement Strategies; Enrollment Flyer & Testimonial Booklet
Other: Teacher Endorsement — Brief conversation between the parent and their child's teacher in which the teacher told the parent about the benefits of participating in the Triple P Positive Parenting Program and recommended that the parent attend. The teacher also gave the parent a brochure that gave information about the Triple P program and an enrollment form.
  Arms: All Engagement Strategies; Enrollment Flyer & Teacher Endorsement
Other: Provider Engagement Call — This was a manualized, 15-minute call from the Triple P Positive Parenting Program provider to a parent in which the provider elicited the parent's child-focused goals and showed how the parent's goals could be addressed by Triple P. The provider also helped the parent anticipate and problem solve possible barriers to attendance.
  Arms: All Engagement Strategies; Enrollment Flyer & Engagement Call

SUMMARY:
This study tests the effectiveness of different strategies for engaging parents into an evidence-based parenting skills intervention, the Triple P Positive Parenting Program, offered universally to parents of children attending one of six public elementary schools.

DETAILED DESCRIPTION:
Parenting skills programs have been shown to help prevent youth substance use and mental health disorders. Unfortunately, few parents participate in parenting programs when given the opportunity. Thus, developing effective strategies to increase engagement in effective preventive parenting interventions is essential for these programs to have a significant public health impact. The purpose of this study is to identify parent engagement strategies that increase participation in effective parenting programs and consequently improve parenting practices and children's well-being.

ELIGIBILITY:
Inclusion Criteria:

* Is a caregiver of a child in kindergarten, 1st, 2nd or 3rd grade at a participating school (i.e.,"target child");
* The target child lives with the caregiver at least half of the time;
* The caregiver speaks English or Spanish;
* The caregiver is listed as one of the target child's parents/guardians in the school's records.

Exclusion Criteria:

* The target child is in a self-contained classroom due to cognitive or emotional disabilities;
* The caregiver is a kindergarten, 1st, 2nd or 3rd grade teacher at a participating school;
* The target child attended one of the participating schools during a previous cohort of the study;
* The caregiver is participating in a competing parenting program at the school, the "Intensive Family Literacy program".

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 854 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Parenting Intervention Attendance | Attendance at the Triple P Positive Parenting Program was collected once per week for 8 weeks
  Number of sessions a caregiver from a student's family attended the parenting intervention, the Triple P Positive Parenting Program

SECONDARY OUTCOMES:
Parenting Intervention Enrollment | from the date engagement strategies commenced until the date the Triple P Positive Parenting Program began, up to 7 weeks
  Whether or not a family enrolled in the Triple P Positive Parenting Program by completing an enrollment form.
Parenting Intervention Homework Completion | collected once per week for 7 weeks, at the beginning of each Triple P Positive Parenting Program sessions 2 through 8
  caregiver report of completion of Triple P Positive Parenting Program assignments between sessions
Parenting Intervention Session Involvement | collected once per week for 8 weeks, after each Triple P Positive Parenting Program session
  group leader reports of the extent to which a caregiver actively participated in each Triple P Positive Parenting Program session attended
Child Behavior Problems | collected at baseline and at Triple P post-test, an average of 7 months after baseline
  parent and teacher reports of child behavior problem frequency and intensity
Parenting Skills | collected at baseline and at Triple P post-test, an average of 7 months after baseline
  parent report of parenting warmth and discipline

CONTACTS AND LOCATIONS:
Overall Officials: Emily B Winslow, Ph.D., Principal Investigator — Arizona State University
Locations (1):
- Arizona State University, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: No